CLINICAL TRIAL: NCT01742624
Title: Multicenter, Open-label, Parallel Clinical Investigation of the Safety and Efficacy of Advagraf® (Extended Release Tacrolimus) vs. Prograf® (Tacrolimus) in de Novo Kidney Recipients 1 Month After Kidney Transplantation
Brief Title: Study to Evaluate the Safety and Efficacy of Advagraf vs Prograf in Kidney Transplantation Patients 1 Month After the Transplantation
Acronym: AdProCISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADV-KT-01
Record Dates: First submitted 2012-12-04; First posted 2012-12-05 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: de Novo Kidney Transplantation
Keywords: immunosuppressant; new-onset diabetes after kidney transplantation; NODAT
MeSH Terms: interventions — Tacrolimus; Adrenal Cortex Hormones; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advagraf group (Experimental)
  Interventions: Drug: Advagraf; Drug: Corticosteroid; Drug: Mycophenolate mofetil
- Prograf group (Active Comparator)
  Interventions: Drug: Prograf; Drug: Corticosteroid; Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Advagraf — oral
  Other Names: tacrolimus
  Arms: Advagraf group
Drug: Prograf — oral
  Other Names: tacrolimus, FK506
  Arms: Prograf group
Drug: Corticosteroid — oral
Drug: Mycophenolate mofetil — oral

SUMMARY:
To investigate the efficacy, safety, and drug compliance of Advagraf® (Extended Release Tacrolimus) by comparing the Advagraf® + steroid + Mycophenolate Mofetil combined therapy and the Prograf® + steroid + Mycophenolate Mofetil combined therapy in de novo kidney recipients 1 month after kidney transplantation.

DETAILED DESCRIPTION:
This study is a multicenter, open-label, randomized, parallel, and comparative clinical trial. All the enrolled subjects will be treated with Prograf® (Tacrolimus), Basilixumab, Corticosteroids, and Mycophenolate Mofetil to suppress their immune system for one month (30 days) after their kidney transplant. After the one month, the experimental group (30 subjects) will be treated with Advagraf® (Extended Release Tacrolimus) instead of Prograf® (Tacrolimus), and the Corticosteroids and Mycophenolate Mofetil will be maintained. The control group (30 subjects) will continuously receive Prograf® (Tacrolimus), Corticosteroids, and Mycophenolate Mofetil. The clinical progress of the subjects in the experimental and control groups up to six months after their transplant will be investigated and compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planning to receive a kidney from a deceased/cadaveric donor or a living non-related/related donor
* Patients who are planning to undergo kidney transplantation through a 15- 65-year-old donor
* Patients who are willing and able to participate in this study, who signed the informed consent form after following the appropriate informed consent process, and who can visit the center based on the study schedule in the protocol.

Exclusion Criteria:

* Patients who had received a kidney or another organ and who will receive other organs with the kidney or two kidneys
* Patients who will receive a kidney from a cadaveric donor whose heart is no longer beating or from an organ donor after cardiac death [Patients, however, who will receive a kidney from a marginal donor (based on KONOS) can be enrolled based on the principal investigator's judgment.]
* Patients who will receive a kidney from a donor whose ABO blood type is not compatible with that of the recipient or who had positive lymphocyte cross-match (LCM) results
* Patients who will receive a kidney from a related donor who showed HLA-0 mismatch (identical) (If the donor is not related to the patient or is deceased, however, the patient can be enrolled in this study even if the patient showed HLA-0 mismatch or HLA-6 antigen match.)
* Patients who previously underwent or are planning to undergo transplantation of their extra-renal solid organ or bone marrow/stem cell
* Patients who were diagnosed with cancer in the last five years [ Patients, however, who have recovered from skin cancer (squamous cell/basal cell carcinoma) can be enrolled.]
* Patients or donors who have positive HIV, HBsAg, or anti-HCV test results
* Patients who have a history of hypersensitivity or allergy [that required acute (within four weeks)/chronic treatment] to the investigated drug or another drug with a similar chemical structure (e.g., Tacrolimus).
* Patients who were treated with other investigated drugs within 30 days from their study enrollment
* Patients who are planning to be pregnant, or who are pregnant or breastfeeding and who are not planning to use any contraceptive method during the study period.
* Patients who were addicted to drugs/alcohol within six months of their study enrollment or who have a mental illness that makes appropriate communication with them impossible
* Patients who showed the following result in the assessment prior to the kidney transplantation

  * Any of their liver panels (AST, ALT, ALKP, and total bilirubin) three times higher than the normal range
  * Absolute neutrophil count < 1,500/mm3, leukocytes < 2,500/mm3, or platelet < 100,000/mm3

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Incidence of efficacy failure (treated-BCAR, biopsy-confirmed acute rejection, graft loss rate, death, or follow-up failure) | until 6 months

SECONDARY OUTCOMES:
Survival rate | at 6 months after treatment
Kidney function (eGFR) | at 6 months
  assessment of eGFR using the Nankivell method
24-hour urine protein and creatinine clearance rate(CCR) | at 6 months
Incidence of new-onset diabetes after kidney transplantation (NODAT) | until 6 months
Safety assessed by the incidence of adverse events, physical exam, and labo-tests | until 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (3):
- South Korea (3):
  - Seoul
  - Suwon
  - Ulsan

REFERENCES:
- [Derived] Oh CK, Huh KH, Lee JS, Cho HR, Kim YS. Safety and efficacy of conversion from twice-daily tacrolimus to once-daily tacrolimus one month after transplantation: randomized controlled trial in adult renal transplantation. Yonsei Med J. 2014 Sep;55(5):1341-7. doi: 10.3349/ymj.2014.55.5.1341. PMID 25048494